CLINICAL TRIAL: NCT03114865
Title: A Phase IB/II Study of Blinatumomab in Patients With Pre B-cell Acute Lymphoblastic Leukemia (ALL) and B-cell Non-Hodgkin Lymphoma (NHL) as Post-allogeneic Stem Cell Transplant (Allo-HSCT) Remission Maintenance
Brief Title: A Study of Blinatumomab in Patients With Pre B-cell ALL and B-cell NHL as Post-allo-HSCT Remission Maintenance
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1713; IRB00125679 (Other: JHMIRB)
Record Dates: First submitted 2017-04-11; First posted 2017-04-14 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Acute Lymphoblastic Leukemia; B-cell Non Hodgkin Lymphoma; Pre B-Cell Acute Lymphoblastic Leukaemia
Keywords: bone marrow; bone marrow transplant; allogeneic; tacrolimus; cyclophosphamide; Blinatumomab
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, B-Cell; Precursor B-Cell Lymphoblastic Leukemia-Lymphoma | interventions — blinatumomab; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Post-alloHSCT Maintenance (Experimental): Blinatumomab will be administered as a continuous intravenous (IV) infusion over four weeks followed by a two-week treatment free interval. It is recommended that patients are hospitalized at least during the first three days of the first cycle and the first two days of the second cycles.
  Interventions: Drug: Blinatumomab 9ug; Drug: Blinatumomab 28 ug; Drug: Blinatumomab; Drug: Dexamethasone

INTERVENTIONS:
Drug: Blinatumomab 9ug — Cycle 1 - Days 1-7: 9 ug/day IV daily
  Other Names: Blincyto
Drug: Blinatumomab 28 ug — Cycle 1 - Days 8-28: 28 ug/day IV daily
  Other Names: Blincyto
Drug: Blinatumomab — Cycle 2 - Days 1-28: 28 ug/day IV daily
  Other Names: Blincyto
Drug: Dexamethasone — Day 1 of Cycle 1 and 2, prior to a step dose (such as cycle 1 day 8), or when restarting an infusion after an interruption of 4 hours or more: 20 mg IV

SUMMARY:
The investigators primary objective is to determine the safety and toxicity of incorporating blinatumomab into the post-allogeneic hematopoietic stem cell transplant (HSCT) maintenance setting for patients with CD19+-B-cell malignancies (Acute Lymphoblastic Leukemia [ALL], Non-Hodgkin's Lymphoma [NHL]).

ELIGIBILITY:
Inclusion Criteria

1. Pre-B ALL, low and high grade NHL who underwent an alloHSCT using posttransplant CY GVHD prophylaxis (Pt-Cy alone or combination with MMF/tacrolimus or sirolimus) as follows:

   A. Pre-B ALL patients in CR1 with high-risk features such as adverse cytogenetics including t(9;22) or Ph-like ALL, t(4;11) or other MLL (KMT2A) rearrangements, t(v;14q23)/IgH, complex karyotype (≥5 chromosomal abnormalities), hypodiploidy (<44 chromosomes), low hypodiploidy (30-39 chromosomes)/near triploidy (60-68 chromosomes), intrachromosomal amplification of chromosome 21 (iAMP21), high WBC count at presentation (≥30,000), lack of achievement of complete remission after standard induction chemotherapy (but achieved CR1 following salvage or consolidation), or persistence of detectable disease after induction and consolidation (intensification) or pre-transplant as documented on any of routine clinical tests (morphology, flow cytometry, cytogenetics or molecular studies) OR all Pre-B ALL patients in second and higher CR B. Low and high grade NHL following a nonmyeloablative (reduced-intensity conditioning) transplant irrespective of pre-transplant disease status
2. Patients should be at least 60 but not more than 180 days from transplant with documented count recovery (ANC >1 x109/L, and non-transfused platelets >30x109/L) and no evidence of disease progression
3. ECOG performance status 0-2
4. Ability to give informed consent
5. In agreement to use an effective barrier method of birth control (hormonal or barrier method of birth control; abstinence) to avoid pregnancy during the study and for a minimum of 30 days after study treatment, for all male and female patients who are fertile
6. Age ≥18 years
7. Patients may have received any number of prior regimens to achieve remission. Patients previously treated with blinatumomab will be eligible as long as they did not experience unacceptable toxicities with prior blinatumomab administration. If patient was refractory (no response) to blinatumomab in the past, patient will be eligible if there was no evidence of CD19 loss on leukemia cells.

Exclusion Criteria

1. Lack of engraftment (less than 85% donor DNA in bone marrow or peripheral blood after allogeneic HSCT).
2. Active or untreated disease in central nervous system or testes
3. Patient has received chemotherapy or radiotherapy (with the exception of intrathecal chemotherapy) within 2 weeks of starting blinatumomab. Patient could receive intrathecal prophylactic chemotherapy within a week prior to starting blinatumomab.
4. Patients with active uncontrolled infection or uncontrolled intercurrent illness including, but not limited to symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
5. Patients with prior history of severe (grade 3 or 4) acute GVHD or active severe chronic GVHD even if resolved will not be eligible. Patients with history of active acute GVHD (grade 2) and active moderate chronic GVHD who required steroids for the treatment of GVHD will need to be off steroids for at least 4 weeks prior to treatment start. (Topical steroids or physiologic adrenal replacement steroid doses are allowed).
6. Patients requiring calcineurin inhibitors (i.e. tacrolimus or sirolimus) or other systemic immunosuppressants (cyclosporine (CNI); methotrexate or similar) for GVHD prophylaxis or treatment within 4 weeks prior to treatment start.
7. Inadequate end organ function defined as AST, ALT, and alkaline phosphatase > 3X ULN, bilirubin >=1.5X ULN, or creatinine >=2 mg/dL
8. Patients with Ph-positive ALL who are eligible for post-transplant TKI maintenance based on a demonstrated sensitivity to TKIs pre-transplant (patients with known intolerance or resistance to TKI will be eligible)
9. Evidence of progressive disease post-transplant
10. Women who are pregnant or lactating
11. Known hypersensitivity to blinatumomab
12. Patients with a concurrent active malignancy for which they are receiving treatment
13. Concurrent use of any other investigational drugs
14. Patient who have a history or presence of clinically relevant CNS pathology such as epilepsy, seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, psychosis, or other significant CNS abnormalities. A history of treated CNS leukemia or lymphoma will be allowed if recent imaging and CSF studies confirm the absence of active CNS disease at the time of study entry
15. Weight <45 kg
16. Patients receiving other post-transplant maintenance therapies
17. Infection with human immunodeficiency virus (HIV) or chronic infection with hepatitis B virus or hepatitis C virus (HCV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival at two years post first treatment cycle | 2 years
  Percentage of enrolled participants who receive BMT and Blinatumomab and are alive at two years post BMT.

SECONDARY OUTCOMES:
Non-Relapse Mortality | 2 years
  Percentage of participants who experience non-relapse mortality after 2 years.
Progression-free survival | 2 years
  Percentage of participants who experience progression-free survival after 2 years.
Disease-free Survival | 2 years
  Percentage of participants who experience disease-free survival after 2 years.
Overall Survival | 2 years
  Percentage of participants who experience overall survival after 2 years.
Minimal Residual Disease | 2 years
  Percentage of participants who convert from MRD to no MRD after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ivana Gojo, MD, Study Chair — Johns Hopkins University; Jonathan Webster, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No